CLINICAL TRIAL: NCT03368794
Title: Naloxone to TReatment Entry in the Emergency Setting
Acronym: N-TREE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Practical difficulties in starting active recruitment.
Sponsor: Anders C Håkansson (Other)
Responsible Party: Sponsor-Investigator, Anders C Håkansson, MD, PhD, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-TREE
Record Dates: First submitted 2017-07-25; First posted 2017-12-11 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Opioid Dependence; Opioid Intoxication; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Telephone alert signal from ambulance staff to out-patient substance use disorder treatment facility, for active outreach aiming to locate and include the patient in long-term evidence-based treatment for the substance use disorder.
  Interventions: Behavioral: Active treatment referral of opioid overdose survivors to long-term treatment
- Control (Active Comparator): Information-only. Ambulance staff hand over written information to the individual about how to seek treatment for the substance use disorder.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Active treatment referral of opioid overdose survivors to long-term treatment — Telephone alert and outreach for inclusion, assessment and intake into long-term evidence-based treatment of the substance use disorder.
  Arms: Intervention
Behavioral: Control — Written information from ambulance staff to the patient about how to seek treatment. Patient is able to contact the research treatment facility through a specific phone number, making it possible to study treatment entry in the information-only control condition.
  Other Names: Information-only
  Arms: Control

SUMMARY:
The study tests a structured referral process for opioid overdose survivors, from pre-hospital emergency care to long-term treatment of the individual's substance use-related disorder.

DETAILED DESCRIPTION:
Randomized controlled trial. Subjects are included if they are being treated by an ambulance in the Malmö uptake are for an opioid overdose requiring naloxone antidote administration, and if they sign informed written consent to the study. Subjects are randomized by ambulance staff to either an active intervention, or a control condition:

Intervention: A telephone alert signal is sent from ambulance staff after successful naloxone reversal of an opioid overdose, leading to an active outreach effort from the staff of the addiction research facility, where staff locate the individual and offer her/him formal inclusion in the study.

Control: No telephone alert signal is sent, and the active outreach procedure is not carried out. Ambulance staff hand over written information to the individual about how she/he can apply actively for treatment.

Primary outcome is entry into formal assessment and treatment of the substance use disorder.

ELIGIBILITY:
Inclusion Criteria:

* survivor of opioid overdose requiring antidote naloxone administration by ambulance staff, and provision of written informed consent

Exclusion Criteria:

* patients unable to understand study information and to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Treatment entry | Two weeks
  Entry into formal assessment for evidence-based treatment of opioid use disorder

SECONDARY OUTCOMES:
Treatment retention | 3, 6, 12, 24 and 36 months
  Retention in opioid maintenance treatment or other relevant evidence-based treatment for the substance-related condition, as measured in treatment records, and including the analysis of predictors of retention
Treatment outcome (urinalysis) | 3, 6, 12, 24 and 36 months
  Drug-free status in treatment, as documented from hospital records of drug-free urines
Treatment outcome (hair analysis) | 3 months
  Drug-free status in treatment, as documented by hair analysis
Treatment outcome (self-report) | 3, 6, 12, 24 and 36 months
  Drug-free status in treatment, described through self-report (AUDIT, DUDIT)
Treatment outcome (quality of life) | 3, 6, 12, 24 and 36 months
  Self-report, EQ-5D (European Quality of life - 5 Dimensions) and visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Anders Håkansson, MD, PhD, Principal Investigator — Lund University. Region Skåne.
Locations (1):
- Malmö Addiction Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No